CLINICAL TRIAL: NCT05048511
Title: Evaluation of the Impact of Vitamine D Status on in Vitro Fertilization Outcomes in a Large Population of Infertile Women.
Brief Title: Impact of Vitamine D Status on in Vitro Fertilization Outcomes
Acronym: DFIV
Status: Withdrawn | Type: Observational
Why Stopped: The project was abandoned because of a lot of publications on the subject in the meantime and it was not considered relevant to continue.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0122
Record Dates: First submitted 2016-05-09; First posted 2021-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Infertility
Keywords: Vitamin D, 25(OH)D; in vitro fertilization; AMH; infertility; clinical pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Women with sufficient vitamin D level, when 25(OH)D >20 ng/ml
  Interventions: Biological: vitamin D estimation
- Deficient: women deficiency vitamin D level, when 25(OH)D <20 ng/ml
  Interventions: Biological: vitamin D estimation

INTERVENTIONS:
Biological: vitamin D estimation — Serum samples to estimate vitamin D status were collected on the sixth day of stimulation

SUMMARY:
Non skeletal effect of vitamin D have been the focus of much interest in the past decade. During the last years, special attention has been given to the impact of vitamin D on human reproduction. Its receptor is expressed in most reproductive organs including hypothalamus, pituitary gland, uterus, ovary, mammary gland and the placenta. In vitro experiments suggest that vitamin D would be involved in regulated embryo-implantation. Concerning AMH, vitamin D seems to alters AMH signaling in human granulosa cells although their circulated levels are correlated in lated reproductive aged women. The results of precedents studies about the impact of vitamin D on IVF outcomes remain conflicting The aim of our study was to assess in a large unselected population of infertile women, the impact of vitamin D deficiency on IVF outcome and to examine the relationship between serum vitamin D levels and the ovarian reserve marker AMH.

DETAILED DESCRIPTION:
Vitamin D was measured on the sixth day of stimulation. According to vitamin D level, women were divided into 2 groups (deficiency when 25(OH)D <20 ng/ml and sufficient when 25(OH)D >20 ng/ml).

Pregnancy rates were compared among these two groups after controlling age, BMI, characteristics of ovarian stimulation, number of ovocytes obtains, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI in the center of medical assistance for the procreation of the french hospital of Nantes between september 2010 and may 2011.

Exclusion Criteria:

* Women for who the cycle was interrupted during ovarian stimulation or converted in intrauterine insemination.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: population of infertile women undergoing IVF/ICSI in the center of medical assistance for the procreation of the french hospital of Nantes between september 2010 and may 2011.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Laboratory pregnancy | 4 weeks to 9 month
  Serum HCG was drawn 16 days after ovocyte tapping; Patient had a repeat bHCG drawn 48 hours if they have a positive result from the first bHCG; Clinical pregnancy was defined as ultrasound documentation of fetal heart tones at seven weeks of gestation
Clinical pregnancy | 4 weeks to 9 month
  Serum HCG was drawn 16 days after ovocyte tapping; Patient had a repeat bHCG drawn 48 hours if they have a positive result from the first bHCG; Clinical pregnancy was defined as ultrasound documentation of fetal heart tones at seven weeks of gestation
Live birth | 4 weeks to 9 month
  Serum HCG was drawn 16 days after ovocyte tapping; Patient had a repeat bHCG drawn 48 hours if they have a positive result from the first bHCG; Clinical pregnancy was defined as ultrasound documentation of fetal heart tones at seven weeks of gestation

SECONDARY OUTCOMES:
The relationship between serum vitamin D levels and the ovarian reserve marker AMH | day 3
  Serum AMH was drawn during hormonal examination on third day of natural cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUBOURDIEU, Dr, Principal Investigator — Nantes University Hospital

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Bouillon R, Carmeliet G, Verlinden L, van Etten E, Verstuyf A, Luderer HF, Lieben L, Mathieu C, Demay M. Vitamin D and human health: lessons from vitamin D receptor null mice. Endocr Rev. 2008 Oct;29(6):726-76. doi: 10.1210/er.2008-0004. Epub 2008 Aug 11. PMID 18694980
- [Background] Halloran BP, DeLuca HF. Effect of vitamin D deficiency on fertility and reproductive capacity in the female rat. J Nutr. 1980 Aug;110(8):1573-80. doi: 10.1093/jn/110.8.1573. PMID 7400847
- [Background] Vigano P, Lattuada D, Mangioni S, Ermellino L, Vignali M, Caporizzo E, Panina-Bordignon P, Besozzi M, Di Blasio AM. Cycling and early pregnant endometrium as a site of regulated expression of the vitamin D system. J Mol Endocrinol. 2006 Jun;36(3):415-24. doi: 10.1677/jme.1.01946. PMID 16720713
- [Background] Evans KN, Nguyen L, Chan J, Innes BA, Bulmer JN, Kilby MD, Hewison M. Effects of 25-hydroxyvitamin D3 and 1,25-dihydroxyvitamin D3 on cytokine production by human decidual cells. Biol Reprod. 2006 Dec;75(6):816-22. doi: 10.1095/biolreprod.106.054056. Epub 2006 Sep 6. PMID 16957024
- [Background] Merhi Z, Doswell A, Krebs K, Cipolla M. Vitamin D alters genes involved in follicular development and steroidogenesis in human cumulus granulosa cells. J Clin Endocrinol Metab. 2014 Jun;99(6):E1137-45. doi: 10.1210/jc.2013-4161. Epub 2014 Mar 14. PMID 24628555
- [Background] Grundmann M, von Versen-Hoynck F. Vitamin D - roles in women's reproductive health? Reprod Biol Endocrinol. 2011 Nov 2;9:146. doi: 10.1186/1477-7827-9-146. PMID 22047005